CLINICAL TRIAL: NCT07302048
Title: Impact and Determinants of Success of a Mobile Multidisciplinary Intervention System Specialized in Pain Management for Patients With Moderate to Severe Intellectual Development Disorder, Isolated or Associated With an ASD or Multiple Disability - MoDIDol
Brief Title: Impact and Determinants of Success of a Mobile Multidisciplinary Intervention System Specialized in Pain Management for Patients With Moderate to Severe Intellectual Development Disorder, Isolated or Associated With an ASD or Multiple Disability
Acronym: MoDIDol
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: Fondation de France (Other); Université de Bretagne Occidentale, Brest-France (Unknown); Fondation Perce Neige (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 29BRC24.0282
Record Dates: First submitted 2025-07-03; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Autism Disorder; Multiple Disabilities; Pain; Intellectual Developmental Disorder
Keywords: Pain; Children; Adolescents; young adults; Intellectual Developmental Disability; Autism Spectrum Disorder; multiple disabilities; mobile team
MeSH Terms: conditions — Autistic Disorder; Pain; Intellectual Disability; Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: MoDIDol is a monocentric, prospective, non-comparative interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- children or young adults with IDD, ASD or multiple disabilities (Experimental): Single arm study
  Interventions are :
  * parents education for NCCPC and PPP by a pain specialized nurse at T1
  * parents fullfilling of questionnaires à T1, T2 and T3 with study engineer
  Interventions: Procedure: MoDIDol intervention

INTERVENTIONS:
Procedure: MoDIDol intervention — Multidisciplinary mobile intervention system specialising in pain management for patients with moderate to severe intellectual development disorders, isolated or associated with ASD or multiple disabilities.
  Treatment recommendations, pain assessment, training in scales, follow-up consultations every 6 weeks for 6 months, continued if the situation is not resolved, call at 12 months.

SUMMARY:
Pain is described by patients with a Neurodevelopmental Disorder (NDD), including Autism Spectrum Disorder (ASD), Intellectual Development Disorder (IDD) or multiple disabilities, and the family as one of the main associated disorders; its management is also one of the main concerns of families and professionals. At present, there is no validated and tested pain management system in populations facing complex pain situations. In response to the lack of a pain management services, a multi-disciplinary mobile team was set up in September 2022 at the Brest University Hospital (Mobile Pain Handicap Team Intellectual Disability 0-25 years; MoDIDol). This team offers a specific protocol for the assessment and management of pain that takes into account the social and family environment, the living context and the clinical characteristics of patients (children, adolescents and young adults (0-25 years) with IDD, ASD or multiple disabilities). The team includes at least one paediatrician specialising in the assessment and treatment of pain and a nurse, and travels to patients' usual living environments.

DETAILED DESCRIPTION:
The MoDIDol team intervenes at the request of parents or professionals in complex situations involving pain or behavioural problems suggestive of pain, unresolved despite previous treatment. Parents and professionals learn about the MoDIDol team through flyers and information provided by associations and organisations supporting people with disabilities (associations, CRDI, etc.).

Once they are included in the study and after consent has been signed, multidisciplinary follow-up consultations are carried out by the MoDIDol team for pain management (every 6 weeks).

At the same time, three data collection sessions are planned for the participants, 3 months apart. Questionnaires are completed at each point by dedicated study staff. Interviews are conducted at 6-month intervals among a representative sample of professionals and parents.

ELIGIBILITY:
Inclusion Criteria:

* Aged from birth up to 24 years inclusive (i.e., under 25 years old)
* Medical diagnosis of intellectual disability (ID), isolated or associated with autism spectrum disorder (ASD), developmental disorder (DD), or profound multiple disabilities, based on international classification systems (ICD-11 or DSM-5)
* Confirmed probable or definite pain diagnosis, as validated by the MoDIDol team
* PGIC score ≥ 3
* Living in or receiving care in the departments of Finistère, Côtes-d'Armor, or Morbihan
* Written informed consent provided by parents, legal guardians, or holders of parental authority, authorizing data collection for research and publication purposes
* Affiliated with or benefiting from a French national health insurance scheme

Exclusion Criteria:

* More than three places of residence and/or care settings
* Parents or legal guardians who do not have sufficient language or comprehension skills to provide informed consent or complete study questionnaires

Max Age: 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2028-04-20 (Estimated); Study Completion 2028-04-20 (Estimated)

PRIMARY OUTCOMES:
Global Clinical Improvement at 6 months | From baseline to the end of 6 months of treatment with the MoDIDol system, assessed up to 6 months (T3)
  The primary outcome is the patient's global clinical improvement as perceived by family caregivers and/or institutional professionals, using the Patient Global Impression of Change (PGIC) scale after 6 months of care provided by the MoDIDol team. Improvement is defined as a PGIC score of 1 or 2 out of 7. scale from 1 to 7, higher scores mean worse outcome.

SECONDARY OUTCOMES:
Global Clinical Improvement at 3 months | From baseline to the end of 3 months of treatment with the MoDIDoL system, assessed up to 3 months (T2)
  Global clinical improvement of the patient, as reported by caregivers and/or professionals, measured using the Patient Global Impression of Change (PGIC) scale after 3 months of MoDIDol care. Improvement is defined as a PGIC score of or 2 out of 7. Scale from 1 to 7, higher scores mean worse outcome.
Non Communicating Children's Pain Checklist (NCCPC) Pain Intensity Scores at T1, T2, and T3 | Baseline (T1), after 3 months (T2), and 6 months (T3) of treatment with the MoDIDol system.
  Pain intensity will be assessed using the french version of Non Communicating Children's Pain Checklist (NCCPC) scale at baseline (T1), 3 months (T2), and 6 months (T3). The full rating is based on a 90-point scale : 4-point scale (0 : not observed ; 3 : frequently) for 30 behavioral assessments. But some behaviors can be omitted when non applicable (NA). Pain is mild if score is between 6 and 10, and moderate to severe if score is 11 or more.
Pediatric Pain Profile (PPP) Pain Intensity Scores at T1, T2, and T3 | Baseline (T1), after 3 months (T2), and 6 months (T3) of treatment with the MoDIDol system.
  Pain intensity will be assessed using the french version of Pediatric Pain Profile (PPP) scale at baseline (T1), 3 months (T2), and 6 months (T3). 20 behaviors are to be rated from 0 = not at all to 3 = completely. Pain is moderate to severe if score is 14/60 or above.
Non Communicating Children's Pain Checklist (NCCPC) Pain Category Change | Baseline (T1), after 3 months (T2), and 6 months (T3) of treatment with the MoDIDol system
  Patients will be categorized based on the french version of Non Communicating Children's Pain Chlecklist (NCCPC) (<6 : no pain; 6 to10 : mild pain; >10 : moderate to severe pain) scores to evaluate changes in pain category from T1 to T2 and T2 to T3. The full rating is based on a 90-point scale : 4-point scale (0 : not observed ; 3 : frequently) for 30 behavioral assessments. But some behaviors can be omitted when non applicable (NA). Pain is mild if score is between 6 and 10, and moderate to severe if score is 11 or more.
Pediatric Pain Profile Pain Category Change | Baseline (T1), after 3 months (T2), and 6 months (T3) of treatment with the MoDIDol system
  Patients will be categorized based on french version of Pediatric Pain Profile (PPP) (<14; > or =14) scores to evaluate changes in pain category from T1 to T2 and T2 to T3. Twenty behaviors are to be rated from 0 = not at all to 3 = completely. Pain is moderate to severe if score is 14/60 or above.
Non Communicating Children's Pain Checklist (NCCPC) Pain Behavior Profiles | Baseline (T1)
  Behavioral indicators of pain will be documented using the item-based responses from Non Communicating Children's Pain Checklist (NCCPC) scale at T1. The full rating is based on a 90-point scale : 4-point scale (0 : not observed ; 3 : frequently) for 30 behavioral assessments. But some behaviors can be omitted when non applicable (NA). Pain is mild if score is between 6 and 10, and moderate to severe if score is 11 or more.
Pediatric Pain Profile Pain Behavior Profiles | Baseline (T1)
  Behavioral indicators of pain will be documented using the item-based responses from Pediatric Pain Profile (PPP) scale at T1. Behaviours are to be assessed from 0 = not at all to 3 = completely (score from 0 to 60; pain if score > 14).
Behavioral Disturbance Evolution | Baseline (T1), after 3 months (T2), and 6 months (T3) of treatment with the MoDIDol system.
  Frequency (0:never to 4: At least once an hour) and severity (1: mild to 3: severe) of three types of behaviors (self-injurious behaviors, stereotypical behaviors, and aggressive/destructive behaviors) will be assessed with the Behavior Problems Inventory (BPI) scale at T1, T2, and T3.
PedsQL Patient Quality of Life Scores | Baseline (T1), after 3 months (T2), and 6 months (T3) of treatment with the MoDIDol system
  Quality of life will be assessed using Pediatric Quality of Life Inventory (PedsQL) for patients without profound disabilities on a five-point Likert scale (from 0: Never/Bad; to 4: Almost Always/Excellent) for 15 items at T1, T2, and T3.
PolyQoL Patient Quality of Life Scores | Baseline (T1), after 3 months (T2), and 6 months (T3) of treatment with the MoDIDol system
  Quality of life will be assessed using Quality of Life Scale for People with polyhandicap (PolyQoL) for patients with profound multiple disabilities on a five-point Likert scale (from 1: very bad; to 5: very goodt) for 21 items at T1, T2, and T3.
Sleep Quality Scores | Baseline (T1), after 3 months (T2), and 6 months (T3) of treatment with the MoDIDol system
  Sleep disorders will be measured with the Sleep Disturbance Scale for Children (SDSC) scale on a five-point Likert scale (from 1: never; to 5: every day) for 25 items at T1, T2, and T3.
Parental Quality of Life | Baseline (T1), after 3 months (T2), and 6 months (T3) of treatment with the MoDIDol system
  Parental quality of life will be assessed using the World Health Organization Quality of Life (WHOQOL-BREF) across four domains rated on a 5-point Likert scale (score from 1 to 5) for 26 items at T1, T2, and T3.
Parental Stress | Baseline (T1), 3 months (T2), and 6 months (T3)
  Parental stress will be evaluated using the Parenting Stress Index (PSI-4) at T1, T2, and T3. This questionnaire includes 120 items divided in two categories (stressors associated with the child domain, or with de parent domain) rated on a 5-point Likert scale ranging from "strongly disagree" to "strongly agree". The total score of stress is obtained by adding up the results. The higher the value is, the higher the stress.
Determinants of Success | From baseline to the end of 6 months of treatment with the MoDIDol system, assessed up to 6 months (T3)
  Individual (e.g., diagnosis, development level, sensory profile) and environmental (e.g., living environment, type of care) factors will be analyzed in relation to PGIC (Patient Global Impression of Change) score at T3.
Pain Mechanism, Localization, and Etiology | Pain mechanism, location and etiology are determined at T1 but can be revised during the 6 months patient follow up
  Pain causes will be described according to the mechanism (nociceptive, neuropathic, nociplastic), location, and etiology. Patients with intellectual deficiency are not able to describe their pain because of verbal impairment. Qualitative informations are available through parents and professionnal observations. Evaluation is based on physical examination, specialized medical advice (dental, ENT, ...) and additional examinations, such as laboratory or medical imaging, if needed. These description are build at T1 as hypothesis and may be specified depending on developments during treatment.
Analgesic and Behavioral Treatments | From baseline to the end of 3 months (T2) and 6 months (T3) of treatment with the MoDIDol system
  Description of treatments (indication and dosage) for pain and behavior at T2 and T3.
Psychometric Properties of Non Communicating Children's Pain Checklist (NCCPC) Scale | Through study completion, an average of 6 months after baseline.
  Internal consistency and structural validity of the french version of Non Communicating Children's Pain Checklist (NCCPC) (for patients with ASD) scale will be assessed.
Psychometric Properties of Pediaric Pain Profile Scale | Through study completion, an average of 6 months after baseline.
  Internal consistency and structural validity of the french version of Pediatric Pain Profile (PPP) scale will be assessed.
Qualitative Interviews with Parents and Professionals | Baseline (T1) and after 6 months (T3) of treatment with the MoDIDol system
  Impact of MoDIDol will be assessed through semi-structured interviews before (T1) and after (T3) of the intervention. Themes include daily impact of pain, beliefs, use of pain assessment tools, and perceived value of the mobile team

CONTACTS AND LOCATIONS:
Overall Officials: Philippe J LE MOINE, MD, Principal Investigator — CHU de Brest; Amandine DUBOIS, PhD, Study Director — Université de Bretagne Occidentale
Locations (1):
- CHU de Brest - Hôpital Morvan, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.